CLINICAL TRIAL: NCT02669199
Title: Between Umbilical Cord Mesenchymal Stem Cells Sources Sweat Gland Samples of Large Area Skin Wound Injury Patients Before and After the Transplant Center, Open, Random, Own More Controlled Clinical Trials
Brief Title: MSCs Source of Sweat Gland Cells of Large Area Skin Injury Patients Transplant of the Wound
Acronym: MSCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-007
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: MSCs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSCs (Experimental): The main purpose of this test is to assess the umbilical cord MSCs between source sample sweat gland cells wound transplanted effectiveness and safety for the treatment of large area skin lesions of the subjects
  Interventions: Biological: MSCs

INTERVENTIONS:
Biological: MSCs — The main purpose of this test is to assess the umbilical cord MSCs between source sample sweat gland cells wound transplanted effectiveness and safety for the treatment of large area skin lesions of the subjects

SUMMARY:
The main purpose of this test is to assess the umbilical cord mesenchymal stem cells (MSCs) UC between source sample sweat gland cells wound transplanted effectiveness and safety for the treatment of large area skin lesions of the subjects

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form when the age of 18 and 60 years old or less or more men or women (not pregnancy) The burned area: 10-20% TBSA, can satisfy the self control Time: early for skin grafts For location: limbs, chest and back

Exclusion Criteria:

* Serious allergic constitution; Have influence on the speed of wound healing of chronic disease patients; According to the researcher's judgment, may endanger the safety of the subjects or scheme compliance of any chronic disease or severe disease, including cancer, severe heart disease, kidney disease, liver disease, respiratory disease, nerve diseases of the nervous system, blood system diseases, etc.; Clinical researchers or for other reasons can't cooperate with the doctors, and other information is not suitable for clinical study of patients.

Can not meet the requirement of the long-term follow-up of patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 12 months
  Frequency and severity of Adverse Events

SECONDARY OUTCOMES:
Relative Wound Area Regression of 40% or More at 12 Week | 12 Week

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing Fu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China